CLINICAL TRIAL: NCT03092596
Title: A Structural Intervention to Improve Substance Abuse Diagnosis and Treatment Practices in HIV Clinic Settings
Brief Title: Integrated Care (iCare) at Mount Sinai to Improve Substance Use Diagnosis and Treatment Practices in HIV Clinic Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ana Ventuneac, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-2634; R01DA041072 (NIH)
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Substance Abuse
Keywords: HIV infection; drug abuse; substance use; alcohol abuse; screening; treatment; primary care; motivational interviewing
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patient-administered screening tool (Experimental): Patients will complete a screener for alcohol and drug misuse.
  Interventions: Behavioral: Patient-administered screening tool
- Patient health navigator-administered screening tool (Experimental): Patient health navigators will administer a screener for alcohol and drug misuse to patients.
  Interventions: Behavioral: Patient health navigator-administered screening tool
- Patient health navigator-assisted linkage to treatment (Experimental): Patient health navigators will be trained in motivational interviewing to engage patients about linkage to substance abuse treatment.
  Interventions: Behavioral: Patient health navigator-assisted linkage to treatment
- Treatment as usual (No Intervention): Patients will receive standard care.

INTERVENTIONS:
Behavioral: Patient-administered screening tool — screener for drug and alcohol misuse - NIDA Quick Screen combined with AUDIT and DAST
  Arms: Patient-administered screening tool
Behavioral: Patient health navigator-administered screening tool — patient health navigator-administered screener
  Arms: Patient health navigator-administered screening tool
Behavioral: Patient health navigator-assisted linkage to treatment — patient health navigator-assisted linkage to substance abuse treatment
  Arms: Patient health navigator-assisted linkage to treatment

SUMMARY:
Substance abuse and dependence is highly prevalent among people living with HIV and significantly exacerbates morbidity and mortality and accelerates HIV disease progression. Antiretroviral therapy (ART) has been the single most important treatment for slowing disease progression. ART adherence and HIV primary care are affected by a complex array of factors in the context of lives impacted by socioeconomic, psychological, and health challenges. Drugs and alcohol play a major role in non-adherence, engagement in care, and poor health outcomes among HIV-infected persons. While evidence is unequivocal that substance use treatment improves health outcomes, systems of care for the detection and treatment of substance abuse and dependence remain fragmented. Integrated approaches are key to the delivery of optimal care. Pragmatic or effectiveness trials can provide the best evidence about clinical practice to inform practitioners and policy makes about the most clinically and cost effective treatment to inform dissemination on a wider scale at the organizational and public health levels. The goal of this trial is to develop and test a comprehensive, integrated program to detect and reduce substance abuse and in turn, to improve ART adherence and HIV, substance use and associated health outcomes among HIV-infected patients. This trial will test the effectiveness of the intervention using a stepped wedge trial design to sequentially implement a screening tool and training of patient health navigators at HIV clinics in NYC.

DETAILED DESCRIPTION:
The goal of this research study is to develop an organizational-level intervention to enhance the adoption of screening for and treatment of substance use disorders among HIV-positive patients receiving care at the Institute for Advanced Medicine HIV primary care clinics. The primary research question is: What is the impact of a brief substance abuse screener and treatment referral process on substance use and HIV-related health outcomes among HIV-infected patients attending HIV care clinics?

The study team will achieve four specific aims:

Aim 1: Develop an intervention to integrate substance abuse treatment with HIV care in a consortium of HIV clinics in New York City. The principal investigator will conduct formative research and utilize the study team's findings about existing systems and approaches utilized at the Mount Sinai Health System to: 1) incorporate a brief screening tool to identify patients in need of further assessment or treatment for substance abuse; and 2) train patient health navigators (PHNs) in motivational interviewing (MI) to engage patients for substance abuse treatment.

Aim 2: Test the effectiveness of the intervention using a stepped wedge trial design to sequentially implement a screening tool and training of PHNs at the IAM HIV clinics. The primary goal is to test the effectiveness of intervention components versus treatment as usual (TAU) in identifying HIV infected persons with a substance use disorder and in linking them to substance abuse treatment. Secondary goals include examining the intersection among problematic substance use, HIV medication adherence, and HIV-related and other comorbid conditions.

Aim 3. Develop optimized technologies within the electronic health record (EHR) system used at the HIV clinics and integrate these with existing substance-use treatment mobile applications to retain patients in recovery and relapse prevention. This will specifically entail use of a MyChart mobile patient portal in an Office of the National Coordinator for Health Information Technology (ONC) certified EHRs (Epic, Epic Systems Corporation, Verona, WI). The Affordable Care Act (ACA) and the Health Information Technology for Economic and Clinical Health (HITECH) Act place strong emphasis on the widespread adoption and implementation of EHR systems.

Aim 4: Assess the cost-effectiveness of implementing this organizational-level intervention. In order to enhance the likelihood of widespread implementation, the study team will conduct analyses to assess the cost-effectiveness of implementing the intervention components versus TAU alone.

ELIGIBILITY:
Inclusion Criteria:

* Registered as a patient at the Institute for Advanced Medicine at Mount Sinai
* 18 years of age or older
* HIV-infected
* Report alcohol use at hazardous levels or drug use in the past year
* Ability to provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3358 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Substance Abuse Diagnosis | 6 months post intervention
  Proportion of patients with an alcohol or drug use diagnosis at each HIV clinic compared to proportion of patients who enroll in substance use treatment
Linkage to Substance Abuse Treatment | 6 months post intervention
  Proportion of patients at each HIV clinic who enroll in substance use treatment

SECONDARY OUTCOMES:
HIV Viral Load | 6 months post intervention
  HIV-related outcomes - HIV RNA
CD4 Cell Count | 6 months post intervention
  HIV-related outcomes - CD4 cell count
Comorbidities | 6 months post intervention
  Number of other health indicators and comorbidities related to heart disease, diabetes mellitus, kidney disease, liver disease, osteoporosis, malignancies, cognitive disorders and chronic obstructive pulmonary disease

CONTACTS AND LOCATIONS:
Overall Officials: Ana Ventuneac, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided